CLINICAL TRIAL: NCT03195244
Title: Aquatic Therapy and Autism Spectrum Disorders
Acronym: AT&ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sloan W. Rush, MD (Other)
Responsible Party: Sponsor-Investigator, Sloan W. Rush, MD, MD, Panhandle Eye Group, LLP
Organization: Panhandle Eye Group, LLP (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AT&ASD
Record Dates: First submitted 2017-06-12; First posted 2017-06-22 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Autism Spectrum Disorder
Keywords: aquatic therapy, hydrotherapy
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Observation (No Intervention)
- One-on-one Aquatic Therapy (Active Comparator)
  Interventions: Other: Aquatic Physical Therapy
- Group Aquatic Therapy (Experimental)
  Interventions: Other: Aquatic Physical Therapy

INTERVENTIONS:
Other: Aquatic Physical Therapy — Swim Whisperer's Aquatic Therapy Sessions
  Arms: Group Aquatic Therapy; One-on-one Aquatic Therapy

SUMMARY:
To compare the efficacy of one-on-one versus group-based aquatic therapy on the social interactions, behaviors and physical activities of children with autism spectrum disorders (ASDs).

ELIGIBILITY:
Eligibility criteria:

* DSM-V diagnosis of Autism Spectrum Disorder or DSM-IV diagnosis of Asperger's syndrome or high functioning atypical autism or pervasive development disorder - not otherwise specified or else the typical clinical findings and suspicion of an ASD
* Treatment naïve to prior aquatic therapy

Exclusion criteria:

* Not willing to undergo an investigational treatment
* Unable to cooperate well enough to safely participate in aquatic therapy under the protocol guidelines
* Known allergies to pool chemicals
* Other significant co-morbidities which may include (but is not limited to): severe cerebral palsy with low motor function, advanced pulmonary disease, home oxygen requirement, spina bifida with low motor function, permanent feeding tubes, poorly controlled seizure disorder, chronic indwelling urinary catheters or any condition causing severe cognitive impairment

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Change in PedsQL Score | Baseline and 10 weeks after intervention
  Survey

CONTACTS AND LOCATIONS:
Locations (1):
- Turn Center, Amarillo, Texas, United States

IPD SHARING:
Plan to Share IPD: No